CLINICAL TRIAL: NCT02693990
Title: A Phase I Trial of Increased Dose Intensity Modulated Proton Therapy (IMPT) for High-Grade Meningiomas
Brief Title: A Trial of Increased Dose Intensity Modulated Proton Therapy (IMPT) for High-Grade Meningiomas
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Helen A. Shih, MD, Attending Radiation Oncologist, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-542; 2U19CA021239-36 (NIH)
Record Dates: First submitted 2016-01-13; First posted 2016-02-29 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Meningioma; Brain Tumor
Keywords: Tumor lining the brain; Meningioma; Brain Tumor
MeSH Terms: conditions — Meningioma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Grade II (Atypical) Meningiomas, STR (Experimental): Patient will be treated at the starting dose of Intensity Modulated Proton Therapy (IMPT) which is pre-determined.
  Interventions: Radiation: Intensity Modulated Proton Therapy (IMPT)
- Grade III (Malignant) Meningiomas, GTR (Experimental): Patient will be treated at a pre determined dose of Intensity Modulated Proton Therapy (IMPT) for the specific cohort.
  Interventions: Radiation: Intensity Modulated Proton Therapy (IMPT)

INTERVENTIONS:
Radiation: Intensity Modulated Proton Therapy (IMPT) — Radiation Therapy - Intensity Modulated Proton Therapy (IMPT)

SUMMARY:
This research study is studying radiation therapy as a possible treatment for meningioma or tumor on the lining of the brain. The study drug or intervention involved in this research study is Intensity Modulated Proton Therapy (IMPT)

DETAILED DESCRIPTION:
This is a Phase I clinical trial. Researchers are trying to find out if using increased-dose intensity modulated proton therapy (IMPT) for treatment of Meningiomas will be more effective than the current treatment.

The intensity modulated part of IMPT allows for even better concentration of the radiation dose to the desired target and less dose to the surrounding normal tissues than even traditional passive scattering proton therapy can do. Proton beams can be regulated to stop within or shortly beyond treatment targets. Therefore there is little exposure of the normal tissue to radiation.

The FDA (the U.S. Food and Drug Administration) has not approved IMPT as a treatment for any disease.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have either:

  * histologically confirmed atypical meningioma, WHO grade II, Simpson grade 4-5 that has been either subtotally resected or biopsied.

OR

* histologically confirmed malignant/anaplastic meningioma, WHO grade III with gross total resection.

In the case of recurrent radiographically gross disease, pathologic diagnosis may be from time of original biopsy and/or surgery. Pathology should be reviewed and confirmed at the Participating Institution.

Patients may or may not have neurofibromatosis type 1 or 2.

* Age 18 years or older.
* ECOG performance status ≤ 2 (Karnofsky Performance Status ≥ 60, see Appendix A)
* The effects of proton radiation therapy on the developing human fetus are known to be teratogenic. For this reason, women of child-bearing potential and all men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of proton therapy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants may not be receiving any other investigational agents.
* Participants may not have received prior cranial irradiation.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or lactating women are excluded from this study because radiation is known to have teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with radiation therapy, breastfeeding should be discontinued if the mother is treated with radiation therapy.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 3 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-02; Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Assess Safety and Utility of Increased Dose IMPT: Dose-limiting toxicity (DLT) using NCI CTC 4.0 | 2 years
  Establish a safe increased-dose of post-operative IMPT with SIB in treating each of two meningioma cohorts: grade II (atypical) with subtotal resection and grade III (malignant) with gross total resection. Dose-limiting toxicity (DLT) using NCI CTC 4.0 will be assessed from the start of protocol treatment. The dose-seeking plan for each meningioma cohort will follow a modified 3+3 design with the starting and reduced doses for CTV and GTV.

SECONDARY OUTCOMES:
The Absence of Progressive or Recurrent Disease | 5 years
  The duration of local tumor control will be measured from the start date of protocol treatment until the date of progressive or recurrent disease or censored at the date of last follow-up for patients still alive with stable disease. The rate of local failure will be estimated separately for each stratum based on the cumulative incidence, with death as a competing risk in the absence of progressive or recurrent disease.
Overall Survival | 2 years
  • Overall survival (OS) will be measured from the start date of protocol treatment until the date of death due to any cause or censored at the date of last follow-up for patients still alive. The rate of OS will be estimated separately for each stratum using the Kaplan-Meier method.
Calculate Linear Energy Transfer Using Computer Simulations Based on the Treatment Plan | 2 years
  • Linear energy transfer (LET) will be plotted against radiographic changes to assess the pattern of their correlation. Graphical methods and descriptive statistics will be used to determine if the relationship may be characterized by a formal model, possibly after data transformation. All strata will be pooled for the analyses of LET and the other physics endpoints, as they are functions of only the radiation physics, not histology or surgery.

OTHER OUTCOMES:
In Vivo Range of the Delivered Proton Pencil-Beams | 2 years
  For a small subset of the treatment fields delivered at MGH, a prompt gamma-ray spectroscopy system will be used to measure gamma-rays that are naturally emitted from proton reactions with the patient. Based on these measurements, the investigators will calculate the position in the patient of the end-of-range of the individual proton pencil-beams. The reproducibility and statistical precision of the calculated end-of-range positions will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Helen A Shih, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas